CLINICAL TRIAL: NCT00984607
Title: Accurate Fluoroscopic Measurement of Adjustable Laparoscopic Gastric Band Stoma Diameter
Brief Title: Measurement of Gastric Band Stoma Diameter
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Raphael Healthcare System (Other)
Responsible Party: Robert Glenn Hayter, II M.D., Hospital of Saint Raphael
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSR-Gastric Band
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2009-09

CONDITIONS: Obesity
Keywords: Laparoscopic Gastric Band; LAP BAND system
MeSH Terms: conditions — Obesity | interventions — Barium Sulfate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- barium sulfate tablet (Experimental): After a standard upper GI evaluation, oral administration of a standard 13 mm barium sulfate tablet was performed and swallowed with dilute liquid barium during fluoroscopic monitoring.
  Interventions: Procedure: barium sulfate tablet

INTERVENTIONS:
Procedure: barium sulfate tablet — After a standard upper GI evaluation, oral administration of a standard 13 mm barium sulfate tablet was performed and swallowed with dilute liquid barium during fluoroscopic monitoring. A spot radiograph was obtained once the barium tablet was in the gastric pouch and the dilute liquid barium was passing through the gastric band stoma.
  Other Names: E-Z-EM, Inc., E-Z-DISK NDC10361-778-01

SUMMARY:
The purpose of this study is to correlate accurate fluoroscopic measurement of gastric band stoma diameter with patient symptoms for optimal band stoma adjustment. Administration of a barium tablet to gastric band patients with dilute liquid barium allows the accurate measurement of the band stoma diameter. The technique is quick, easy to perform, and eliminates magnification error intrinsic to fluoroscopy. The study data suggests the optimal calibrated gastric band stoma diameter is 3.0 mm. The accurate fluoroscopic measurement of gastric band stoma diameter can optimize band stoma adjustment and improve patient outcomes.

DETAILED DESCRIPTION:
Ten patients presenting for an upper GI series with laparoscopically placed gastric bands were enrolled after informed consent. After a standard upper GI evaluation, oral administration of a standard 13 mm barium sulfate tablet was performed and swallowed with dilute liquid barium during fluoroscopic monitoring. A spot radiograph was obtained once the barium tablet was in the gastric pouch and the dilute liquid barium was passing through the gastric band stoma. Post-processing software used the longest radiographic dimension of the 13 mm barium tablet as the size reference to calibrate measurement of the gastric band stoma diameter.

ELIGIBILITY:
Inclusion Criteria:

* eating
* s/p LAP BAND placement

Exclusion Criteria:

* immediately post operative
* s/p LAP BAND placement
* significant abnormality found on preceding standard upper GI series

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Correlate accurate fluoroscopic measurement of gastric band stoma diameter with patient symptoms for optimal band stoma adjustment. | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Hayter, MD, Principal Investigator — Hospital of Saint Raphael
Locations (1):
- Hospital of Saint Raphael, New Haven, Connecticut, United States